CLINICAL TRIAL: NCT02224976
Title: Impact of Intense Exercise Training on Energy Availability, Ovarian Function and Bone Turnover in Female Athletes
Brief Title: Effect of Intense Training on Ovarian Function and Bone Turnover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FL94
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-09

CONDITIONS: Amenorrhea
Keywords: exercise training
MeSH Terms: conditions — Amenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensified training (Experimental): Volunteers will increase exercise training by 30% from baseline
  Interventions: Behavioral: Intensified Training

INTERVENTIONS:
Behavioral: Intensified Training — Volunteers will increase exercise training by 30% from baseline

SUMMARY:
The investigators propose a prospective, longitudinal, department funded study protocol to evaluate whether changes in energy availability, during a period of highly intensified exercise training, will increase bone turnover markers and decrease ovarian function and exercise performance, in a dose-dependent fashion in competitive female athletes.

DETAILED DESCRIPTION:
Female athletes participating in sports which emphasize leanness as a factor to success, while also imposing large exercise training loads, present a high prevalence of endocrine and metabolic alterations linked to low energy stores, including suppressed ovarian function and bone loss. Increased bone turnover resulting from low energy stores and suppressed estrogen production may hold the most adverse consequences for long term health, increasing the risk of premature osteopenia, while increasing the risk of stress fractures in the short term. Chronically low energy stores may also contribute to the development of overreaching and overtraining syndromes, characterized by excessive, lasting fatigue and long-term decreases in performance, which can compromise these athletes' health and athletic career. The investigators propose the first longitudinal study aiming to demonstrate the link between low energy status, impaired ovarian function, bone turnover and decreased performance in free-living, competitive female athletes. After a 4-week baseline period of habitual training, athletes will undergo 4 weeks of intensified training (IT), during which the exercise load is increased by 30% from their individual baseline load in order to sharply increase energy expenditure. As athletes will be let to freely adjust their food intake, the investigators aim to test the hypothesis that athletes will fail to adjust food intake sufficiently to match energy expenditure, and that the resulting decrease in energy availability (EA, energy intake - energy expenditure from exercise) will influence, in a dose-dependent fashion, the suppression of estrogen production, the increase in bone turnover and the severity of performance decrement. The IT period will then be followed by a 2-week taper (REC), in which exercise training volume will be reduced by 50% from baseline. The investigators will assess whether EA returns to baseline values, and characterize changes in bone turnover during this recovery period. It is hypothesized that any improvements in exercise performance resulting from IT + REC will occur in athletes who were able to remain closest to a balanced energy state during IT. Concretely linking EA to both performance and bone health may incentivize female athletes to adopt more adequate feeding behaviors for their activity level.

ELIGIBILITY:
Inclusion Criteria:

* competitive endurance runners (racing in events ranging from 10km to ultra-marathons)
* training at least 5 days per week over the past 12 months, and more than 30 miles per week
* regular menstrual cycles (24-35 days) over the past 6 months
* maximal oxygen consumption (VO2max) > 50ml/kg/min
* English speaking

Exclusion Criteria:

* smoker
* amenorrhea
* pregnant or lactating in the past 2 years
* chronic disease that will affect bone health, metabolism or the cardiorespiratory system
* take medications that have cardiovascular or metabolic effects
* present any contra-indication to exercise testing (cardiovascular abnormalities)
* report any major illness or injury preventing training for more than 4 weeks over the past 3 months
* a history of clinical anorexia nervosa or bulimia nervosa

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in energy availability (energy intake - energy expenditure of physical activity) | Baseline (week 4), after 4 weeks of intensified training (week 8) and after a two-week recovery period (week 10)
  The investigators aim to capture the spectrum and variability of energy availability in endurance athletes under normal training conditions, describing in detail training regimen, total energy expenditure and nutrition habits during three distinct phases of training that are habitually followed by endurance athletes.

SECONDARY OUTCOMES:
Change in athletic performance | Baseline (week 4), after 4 weeks of intensified training (week 8) and after a two-week recovery period (week 10)
  The investigators will measure the effect of energy availability on exercise performance during baseline, after 4 weeks of intensified training, and after a 2-week recovery, by measuring the relationship of energy availability to maximal oxygen consumption (VO2max) and 3200 meter time trial performance. The investigators will test the hypothesis that performance will be affected by changes in energy availability in a dose-dependent fashion.
Change in ovarian function | Baseline (week 4), after 4 weeks of intensified training (week 8) and after a two-week recovery period (week 10)
  The investigators will measure salivary estradiol and progesterone concentrations daily throughout the study, in order to test the hypothesis that ovarian function may be suppressed by intensified training and decreased energy availability.
Change in bone turnover markers | Baseline (week 4), after 4 weeks of intensified training (week 8) and after a two-week recovery period (week 10)
  The investigators will measure plasma bone turnover markers during baseline and at the end of the intensified training period, in order to test the hypothesis that bone turnover may be compromised by intensified training and decreased energy availability.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen A Casazza, PhD, Principal Investigator — University of California, Davis
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schaal K, VanLoan MD, Hausswirth C, Casazza GA. Decreased energy availability during training overload is associated with non-functional overreaching and suppressed ovarian function in female runners. Appl Physiol Nutr Metab. 2021 Oct;46(10):1179-1188. doi: 10.1139/apnm-2020-0880. Epub 2021 Mar 2. PMID 33651630
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/Main/docs.htm?docid=11240
- See also: UC Davis Sports Medicine — http://www.ucdmc.ucdavis.edu/sportsmedicine